CLINICAL TRIAL: NCT01064440
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of VM202 (Engensis) in Subject With Critical Limb Ischemia
Brief Title: Safety and Efficacy Study Using Gene Therapy for Critical Limb Ischemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMCLI-II-09-002/E
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Critical Limb Ischemia
Keywords: Painful legs; Ischemic legs; Treatment for Claudication; Gene therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose VM202 (Experimental): Patients in this group received 8mg total of VM202. Day 0: 4mg of VM202 (16 injections of 0.5ml of VM202) Day14: 4mg of VM202 (16 injections of 0.5ml of VM202) Day 28: 16 injections of 0.5ml of normal saline Day 42: 16 injections of 0.5ml of normal saline
  Interventions: Biological: Low Dose VM202; Other: Placebo
- High Dose VM202 (Experimental): Patients in this treatment group received a total of 16mg VM202. Day 0: 4mg of VM202 (16 injections of 0.5ml of VM202) Day14: 4mg of VM202 (16 injections of 0.5ml of VM202) Day 28: 4mg of VM202 (16 injections of 0.5ml of VM202) Day42: 4mg of VM202 (16 injections of 0.5ml of VM202)
  Interventions: Biological: High Dose VM202
- Placebo (Sham Comparator): Patients in this group received a total of 8ml normal saline. Day 0: 16 injections of 0.5ml of normal saline Day 14: 16 injections of 0.5ml of normal saline Day 28: 16 injections of 0.5ml of normal saline Day 42: 16 injections of 0.5ml of normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Low Dose VM202 — Day 0: 4mg of VM202 (16 injections of 0.5ml of VM202) Day14: 4mg of VM202 (16 injections of 0.5ml of VM202)
  Other Names: DNA Plasmid; HGF-X7
  Arms: Low Dose VM202
Biological: High Dose VM202 — Day 0: 4mg of VM202 (16 injections of 0.5ml of VM202) Day 14: 4mg of VM202 (16 injections of 0.5ml of VM202) Day 28: 4mg of VM202 (16 injections of 0.5ml of VM202) Day 42: 4mg of VM202 (16 injections of 0.5ml of VM202)
  Other Names: DNA Plasmid; HGF-X7
  Arms: High Dose VM202
Other: Placebo — Day 0: 16 injections of 0.5ml of normal saline Day 14: 16 injections of 0.5ml of normal saline Day 28: 16 injections of 0.5ml of normal saline Day 42: 16 injections of 0.5ml of normal saline
  Other Names: Normal Saline
  Arms: Low Dose VM202; Placebo

SUMMARY:
The purpose of this study is to evaluate whether intramuscular injections of VM202 into the calf is safe and effective in the treatment of critical limb ischemia.

DETAILED DESCRIPTION:
In the absence of revascularization options, most patients with CLI require amputation within 6 months. Patients requiring major amputation face a diminished quality of life, an unfavorable natural history and need extensive resources for their post-amputation rehabilitation and course. The 1-year amputation-free survival rate for patients diagnosed with CLI is 45%; the mortality rate is approximately 25% and may be as high as 45% in those who have undergone amputation. Management of this end-stage disease process consumes a significant amount of healthcare resources. Clearly, new therapeutic approaches are required.

Hepatocyte growth factor (HGF) has been shown to be a potent angiogenic growth factor stimulating the growth of endothelial cells and migration of vascular smooth muscle cells. Because of its pluripotent capabilities, increasing the availability of HGF in ischemic tissues to achieve therapeutic angiogenesis has been a growing area of research.

This study will use VM202, which is a DNA plasmid that contains novel genomic cDNA hybrid human HGF coding sequence (HGF-X7) expressing two isoforms of HGF, HGF 728 and HGF 723. As there are currently no approved drugs that can reverse CLI and as most patients have exhausted surgical and endovascular intervention options, inducing angiogenesis in the affected limb with VM202 may result in an increase in tissue perfusion, which, in turn improve wound healing, reduce pain and improve limb salvage rates.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 90 years of age;
* Diagnosis of critical limb ischemia (Rutherford Class 4 or 5), including:

  * A resting ankle systolic pressure (in either the dorsalis pedis or posterior tibial arteries) of ≤ 70 mmHg in the affected limb; or
  * A resting toe systolic pressure of ≤ 50 mmHg in the affected limb; or
  * For patients in which measurement of ankle systolic pressure is not feasible (e.g. vessel calcification and non-compressibility); TcPO2 ≤ 30 mmHg;
* Poor or suboptimal candidate for bypass graft surgery or percutaneous angioplasty;
* Pain at rest, and/or ischemic ulcers, and/or focal gangrene (< 3 cm2) for a minimum of 2 weeks,
* Significant stenosis (≥ 75%) of one or more of the following arteries: superficial femoral, popliteal, or two or more infra-popliteal arteries as verified by angiography within 12 months prior to enrollment;
* Be willing to maintain current drug therapy for peripheral arterial disease throughout the course of the study including an anti-platelet and statin treatment unless not tolerated;
* Clinically stable on optimized medical regimen for >30 days
* Be capable of understanding and complying with the protocol and signing the informed consent document prior to being subjected to any study related procedures;
* Women who are surgically sterile or at least 1 year postmenopausal or who have been practicing adequate contraception for at least 12 weeks prior to entering the study. If the subject is of child-bearing potential, she must have a negative urine pregnancy test result prior to study enrollment and must agree to repeat pregnancy screening tests during the study. If the subject or the subject's partner(s) is of child bearing potential, the subject and the subject's partner(s) must agree to use a "double barrier" method of birth control while participating in this study.

Exclusion Criteria:

* Subjects who have undergone a successful revascularization procedure or sympathectomy within 12 weeks prior to study entry. A clinically unsuccessful revascularization procedure is defined as one in which:

  * the target vessel re-occludes (≥50%, as verified by a second angiogram. Duplex ultrasonography can be used to determine vessel patency if the patient cannot tolerate a second angiogram), or
  * the target vessel remains patent, but there is no resolution of symptoms 6 weeks after the procedure (e.g. no evidence of ulcer healing, no improvement in pressures, no reduction in resting pain);
* Subjects that will require an amputation in the target leg within 4 weeks of randomization;
* Subjects with evidence of active infection (e.g., cellulitis, osteomyelitis) or deep ulceration exposing bone or tendon in the extremity planned for treatment;
* Heart Failure with a NYHA classification of III or IV;
* Stroke (NIH scale >2) or myocardial infarction within last 3 months;
* Unstable angina
* Uncontrolled hypertension defined as sustained systolic blood pressure (SBP) > 200 mmHg or diastolic BP (DBP) > 110 mmHg at baseline/screening evaluation;
* Ophthalmologic conditions pertinent to proliferative retinopathy or conditions that preclude standard ophthalmologic examination;
* Inflammatory disorder of the blood vessels (inflammatory angiopathy, such as Buerger's disease);
* Subjects with advanced liver disease including decompensated cirrhosis, jaundice, ascites or bleeding varices;
* Subjects currently receiving immunosuppressive medications chemotherapy, or radiation therapy;
* Positive HIV or HTLV at screening;
* Active Hepatitis B or C infection as determined by Hepatitis B surface antibody (HBsAb), Hepatitis B core antibody (IgG and IgM; HBcAb), Hepatitis B surface antigen (HBsAg) and Hepatitis C antibodies (Anti-HCV), at Screening;
* Specific laboratory values at Screening including: Hemoglobin < 8.0 g/dL, WBC < 3,000 cells per microliter, platelet count <75,000/mm3, AST and/or ALT > 3 times the upper limit of normal or any other clinically significant lab abnormality which in the opinion of the investigator should be exclusionary;
* Patients with a recent history (< 5 years) of or new screening finding of malignant neoplasm except basal cell carcinoma or squamous cell carcinoma of the skin (if excised and no evidence of recurrence); patients with family history of colon cancer in any first degree relative are excluded unless they have undergone a colonoscopy in the last 12 months with negative findings;
* Elevated PSA unless prostate cancer has been excluded;
* Subjects with any co- morbid conditions likely to interfere with assessment of safety or efficacy or with an estimated life expectancy of less than 6 months
* Subjects requiring > 81 mg daily of acetylsalicylic acid; If > 81 mg are taken at screening, subjects may be enrolled if willing/able to switch to another medication;
* Subjects requiring regular COX-2 inhibitor drug(s) or high dose steroids (excepting inhaled steroids);
* Major psychiatric disorder in past 6 months;
* History of drug or alcohol abuse / dependence in the past 2 years;
* Use of an investigational drug or treatment in past 12 months; concurrent participation in investigational protocol or unapproved therapeutics and
* Unable or unwilling to give informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-07-09 (Actual); Primary Completion 2013-08-05 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emerson Perin, MD, Principal Investigator — Texas Heart Institute
Locations (16):
- United States (13):
  - Cardiology PC, Birmingham, Alabama
  - Vascular and Interventional Specialist of Orange County, Orange, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Jobst Vascular, Toledo, Ohio
  - University of Oklahoma HSC, Oklahoma City, Oklahoma
  - Texas Heart Institute, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- South Korea (3):
  - Seoul National University, Seoul, Jongno-gu
  - Yonsei University Health System. Severance Cardiovascular Hospital, Seoul, Seodaemun-gu
  - Ewha Womans University Medical Center, Seoul, YangCheon-ku

REFERENCES:
- [Background] Kibbe MR, Hirsch AT, Mendelsohn FO, Davies MG, Pham H, Saucedo J, Marston W, Pyun WB, Min SK, Peterson BG, Comerota A, Choi D, Ballard J, Bartow RA, Losordo DW, Sherman W, Driver V, Perin EC. Safety and efficacy of plasmid DNA expressing two isoforms of hepatocyte growth factor in patients with critical limb ischemia. Gene Ther. 2016 Mar;23(3):306-12. doi: 10.1038/gt.2015.110. Epub 2015 Dec 8. PMID 26649448
- See also: Plasmid DNA of HGF in patients with critical limb ischemia — https://pubmed.ncbi.nlm.nih.gov/26649448/

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Engensis (8 mg): Subjects in this group received 8 mg total of Engensis (VM202) Day 0: 4 mg Engensis (16 injections of 0.5 mL Engensis) Day14: 4 mg Engensis (16 injections of 0.5 mL Engensis) Day 28: 16 injections of 0.5 mL of normal saline Day 42: 16 injections of 0.5 mL of normal saline
  Low Dose VM202: Day 0: 4mg of VM202 (16 injections of 0.5ml of VM202) Day14: 4mg of VM202 (16 injections of 0.5ml of VM202)
  Placebo: Day 0: 16 injections of 0.5ml of normal saline Day 14: 16 injections of 0.5ml of normal saline Day 28: 16 injections of 0.5ml of normal saline Day 42: 16 injections of 0.5ml of normal saline
- High Dose Engensis (16 mg): Subjects in this treatment group received a total of 16 mg Engensis (VM202) Day 0: 4 mg Engensis (16 injections of 0.5 mL Engensis) Day14: 4 mg of Engensis (16 injections of 0.5 mL Engensis) Day 28: 4 mg of Engensis (16 injections of 0.5 mL Engensis) Day42: 4 mg of Engensis (16 injections of 0.5 mL Engensis)
  High Dose Engensis: Day 0: 4 mg Engensis (16 injections of 0.5 mL Engensis) Day 14: 4 mg Engensis (16 injections of 0.5 mL Engensis) Day 28: 4 mg Engensis (16 injections of 0.5 mL Engensis) Day 42: 4 mg Engensis (16 injections of 0.5 mL Engensis)
- Placebo: Subjects in this group will receive a total of 8ml normal saline. Day 0: 16 injections of 0.5 mL of normal saline Day 14: 16 injections of 0.5 mL of normal saline Day 28: 16 injections of 0.5 mL of normal saline Day 42: 16 injections of 0.5 mL of normal saline
  Placebo: Day 0: 16 injections of 0.5 mL of normal saline Day 14: 16 injections of 0.5 mL of normal saline Day 28: 16 injections of 0.5 mL of normal saline Day 42: 16 injections of 0.5 mL of normal saline
Period: Overall Study
Arm/Group | Low Dose Engensis (8 mg) | High Dose Engensis (16 mg) | Placebo
Started | 21 | 20 | 11
Completed | 18 | 17 | 8
Not Completed | 3 | 3 | 3
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Non-compliance | 0 | 1 | 0
Not completed — Death | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Other: amputation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Engensis 8 mg: Subjects in this group received 8 mg total of Engensis (VM202) Day 0: 4 mg Engensis (16 injections of 0.5 mL, 0.25 mg Engensis) Day14: 4 mg Engensis (16 injections of 0.5 mL. 0.25 mg Engensis) Day 28: 16 injections of 0.5 mL of normal saline Day 42: 16 injections of 0.5 mL of normal saline
- Engensis 16 mg: Subjects in this group received a total of 16 mg Engensis (VM202) Day 0: 4 mg Engensis (16 injections of 0.5 mL, 0.25 mg Engensis) Day14: 4 mg of Engensis (16 injections of 0.5 mL, 0.25 mg Engensis) Day 28: 4 mg of Engensis (16 injections of 0.5 mL, 0.25 mg Engensis) Day42: 4 mg of Engensis (16 injections of 0.5 mL, 0.25 mg Engensis)
- Placebo: Subjects in this group received a total of 8 mL normal saline. Day 0: 16 injections of 0.5 mL of normal saline Day 14: 16 injections of 0.5 mL of normal saline Day 28: 16 injections of 0.5 mL of normal saline Day 42: 16 injections of 0.5 mL of normal saline
- Total: Total of all reporting groups
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo | Total
Number analyzed (Participants) | 21 | 20 | 11 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (10.7) | 67.2 (10.9) | 64.3 (14.5) | NA (NA) — The total for AGE was not summarized for the group. It was provided only for each arm. Note this was analyzed in 2013 and is an old study and the analysis cannot be repeated.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 5 | 19
  Male | 14 | 13 | 6 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 7 | 2 | 13
  White | 13 | 11 | 6 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  South Korea | 2 | 1 | 2 | 1
  United States | 19 | 19 | 9 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events Following Intramuscular Administration of 8 and 16 mg Engensis (VM202) or Placebo in Subjects With Critical Limb Ischemia.
Description: The number of participants with treatment-emergent adverse events (TEAEs), defined as adverse events occurring after the first injection of Engensis (VM202), was assessed in moderate or high-risk Critical Limb Ischemia subjects.
Time Frame: Baseline - Days 0, 14, 28, 42, 49, 90, 180, 270 and 365
Population: The Safety Population included all subjects who received at least 1 study drug injection of Engensis or Placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Engensis (8 mg) | High Dose Engensis (16 mg) | Placebo
Number analyzed (Participants) | 21 | 20 | 11
Participants
  Infections and infestations | 8 | 10 | 6
  Cellulitis | 3 | 1 | 1
  Gangrene | 0 | 3 | 2
  Urinary tract infection | 2 | 1 | 2
  Wound infection | 1 | 2 | 0
  Cystitis | 0 | 2 | 0
  Sinusitis | 0 | 2 | 0
  Tooth Abscess | 0 | 0 | 2
  Gastrointestinal disorders | 9 | 7 | 7
  Diarrhoea | 3 | 2 | 2
  Constipation | 2 | 1 | 3
  Nausea | 2 | 2 | 2
  Gastritis | 1 | 2 | 1
  Vomiting | 1 | 1 | 2
  Hiatus hernia | 0 | 2 | 0
  General disorders and administration site conditions | 12 | 6 | 5
  Oedema peripheral | 3 | 2 | 1
  Injection site haematoma | 2 | 0 | 2
  Pyrexia | 0 | 2 | 1
  Musculoskeletal and connective tissue disorders | 9 | 8 | 4
  Pain in extremity | 4 | 6 | 2
  Muscle spasms | 4 | 0 | 1
  Arthralgia | 3 | 1 | 0
  Vascular disorders | 9 | 7 | 4
  Peripheral arterial occlusive disease | 2 | 4 | 1
  Arterial thrombosis limb | 0 | 2 | 0
  Metabolism and nutrition disorders | 5 | 6 | 5
  Hypoglycaemia | 2 | 2 | 2
  Decreased appetite | 0 | 2 | 2
  Hyperglycaemia | 1 | 1 | 2
  Skin and subcutaneous tissue disorders | 8 | 3 | 5
  skin ulcer | 4 | 1 | 2
  blister | 0 | 1 | 2
  Injury, poisoning and procedureal complications | 8 | 3 | 4
  Contusion | 2 | 1 | 2
  Procedural pain | 3 | 1 | 1
  Limb injury | 1 | 2 | 0
  Nervous system disorders | 1 | 7 | 3
  Headache | 0 | 2 | 1
  Phantom pain | 1 | 2 | 0
  Dizziness | 0 | 0 | 2
  Renal and urinary disorders | 7 | 2 | 2
  Renal failure acute | 5 | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 6 | 5 | 0
  Chronic obstructive pulmonary disease | 1 | 2 | 0
  Dyspnoea | 1 | 2 | 0
  Psychiatric disorders | 4 | 5 | 1
  Anxiety | 2 | 2 | 0
  Mental status changes | 1 | 2 | 0
  Depression | 0 | 2 | 0
  Blood and lymphatic system disorders | 5 | 1 | 3
  Anaemia | 4 | 1 | 3
  Cardiac disorders | 3 | 4 | 2
  Acute myocardial infarction | 0 | 2 | 0

2. Primary Outcome: Change From Baseline in Visual Analog Scale (VAS) for Pain
Description: The Visual Analog Scale (VAS) for Pain scoring instrument is a 10 cm line, oriented horizontally, with the left end score of "0" indicating "no pain", and the right end score of "10" representing "pain as bad as it can be"
Time Frame: Days 0, 90, 180, 270, and 365
Population: The Per-Protocol (PP) Population included all subjects who received the correct dose of study drug, had the 9-month (Day 270) VAS assessment, and did not have any protocol violations or major deviations. The PP Population was determined in a blinded review before database lock. Subjects were analyzed according to the treatment to which they were randomized. Primary efficacy analyses were performed on the PP population.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Engensis 8 mg: Subjects received 8 mg total of Engensis Day 0: 4 mg Engensis (16 injections of 0.5 mL, 0.25 mg Engensis) Day14: 4 mg Engensis (16 injections of 0.5 mL, 0.25 mg Engensis) Day 28: 16 injections of 0.5 mL of normal saline Day 42: 16 injections of 0.5 mL of normal saline
- Engensis 16 mg: Subjects received a total of 16 mg Engensis Day 0: 4 mg Engensis (16 injections of 0.5 mL, 0.25 mg Engensis) Day14: 4 mg of Engensis (16 injections of 0.5 mL, 0.25 mg Engensis) Day 28: 4 mg of Engensis (16 injections of 0.5 mL, 0.25 mg Engensis) Day42: 4 mg of Engensis (16 injections of 0.5 mL, 0.25 mg Engensis)
- Placebo: Subjects received a total of 8 mL normal saline. Day 0: 16 injections of 0.5 mL of normal saline Day 14: 16 injections of 0.5 mL of normal saline Day 28: 16 injections of 0.5 mL of normal saline Day 42: 16 injections of 0.5 mL of normal saline
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
Number analyzed (Participants) | 15 | 12 | 5
units on a scale
  Baseline (Day 0) - Actual values only | 40.5 (31.3) | 62.3 (22.5) | 60.6 (30.1)
  Day 90 | -13.0 (15.1) | -32.7 (19.8) | -29.0 (19.9)
  Day 180 | -17.2 (25.6) | -28.9 (31.1) | -29.0 (28.5)
  Day 270 | -8.2 (22.3) | -34.5 (39.6) | -38.6 (41.1)
  Day 365 | -17.6 (30.3) | -29.1 (21.7) | -45.8 (30.8)

3. Secondary Outcome: Change From Baseline in Tissue Oxygenation (TcPO2) for the Dorsal Surface of the Foot Following Engensis (VM202) or Placebo
Description: Tissue Oxygenation (TcPO2) measurement is reported for the dorsum of the foot. The change in baseline for the TcPO2 measured in the dorsal surface of the foot results are reported for each of the 3 study groups: 8 mg, or 16 mg for the Engensis (VM202) group, or the Placebo group. Because of the indication being peripheral vascular disease, the dorsal surface of the foot was decided by the sponsor to be a good representative of the lower extremity for any of the other measured sites.
Time Frame: Day 0 to Days 180, 270, and 365
Population: The Intent-to-Treat population included all subjects who were randomized regardless of whether treatment was received
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 11
mmHg
  Baseline (Day 0) Actual values only | 33.4 (19.4) | 35.0 (18.4) | 40.3 (21.5)
  Day 180: number analyzed (Participants) | 18 | 14 | 6
  Day 180 | 5.9 (19.7) | 7.1 (16.6) | -9.6 (13.5)
  Day 270: number analyzed (Participants) | 18 | 15 | 6
  Day 270 | 3.6 (19.0) | 1.7 (17.8) | -7.1 (14.4)
  Day 365: number analyzed (Participants) | 18 | 15 | 7
  Day 365 | 4.1 (20.5) | 13.4 (15.6) | -9.1 (15.3)

4. Secondary Outcome: Change From Baseline in Hemodynamic Assessment for Ankle Brachial-Index (mmHg) for the Index Leg
Description: Change in the Resting Ankle-Brachial Index (ABI) from Baseline (Day 0) for the Index Leg to Days 180, 270, and 365.
  Note that by default, Day 0 has no change from baseline. Days 28 and 90 time point data was not included,as they were not relevant to assess efficacy, because of the delayed effect of Engensis, the investigational product.
Time Frame: Days 0, 28, 90, 180, 270, and 365
Population: Intent-to-treat population: includes all subjects who were randomized regardless of whether treatment was received
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 11
mm Hg
  Day 180 | 0.009 (0.130) | -0.004 (0.239) | 0.112 (0.267)
  Day 270 | 0.006 (0.181) | 0.010 (0.276) | 0.042 (0.216)
  Day 365 | -0.012 (0.123) | -0.011 (0.277) | -0.010 (0.142)

5. Secondary Outcome: Change From Baseline in Perfusion of the Occluded Target Artery by Magnetic Resonance Angiogram (MRA)
Description: The quantitative blood flow of the occluded target artery and the volumetric analysis of the newly developed artery by Magnetic Resonance Angiogram (MRA) were recorded.
  Note that "no change from baseline table of data" is not presented because there was only one subject with both a Baseline and Post Treatment value for Magnetic Resonance Angiogram (MRA) measurement.
Time Frame: Day 0 to Days 180 and 270
Population: ITT population or Per protocol population - Note: Only 1 subject had both a baseline and post-treatment MRA performed. Unfortunately, no quantitative perfusion data were collected.
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Subjects With 100% Wound Healing
Description: The length and width (in cm) was based on photographs and measurements of ulcers. If a ulcer was determined to be 100% healed, the area of the ulcer was set to 0
Time Frame: Days 0, 14, 28, 42, 49, 90, 180, 270, and 365
Population: Intent-to-Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
Number analyzed (Participants) | 13 | 8 | 4
Participants
  Day 14 | 1 | 3 | 0
  Day 28 | 1 | 4 | 0
  Day 42 | 2 | 4 | 0
  Day 49 | 2 | 4 | 0
  Day 90 | 4 | 4 | 0
  Day 180 | 8 | 4 | 0
  Day 270 | 7 | 3 | 0
  Day 365 | 5 | 3 | 0

7. Secondary Outcome: Change From Baseline in the Vascular Quality of Life Total Score
Description: The Vascular Quality of Life Total Score (VascuQol) questionnaire has 25 questions that reviewed five domains: activity level (8 items), symptoms (4 items), pain (4 items), emotional (7 items), and social (2 items). The total score is the total of the non-missing scored divided by the number of responded questions.
  The Vascular Quality of Life Total Score (VascuQol) scale is a 7-point scale with "1" as the worst change from baseline score, and "7" is the least change from baseline score.
Time Frame: Days 0, 90, 270, and 365
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
Number analyzed (Participants) | 15 | 12 | 5
score on a scale
  Baseline (Day 0) - Actual values only | 3.57 (1.13) | 3.20 (1.15) | 3.50 (1.60)
  Day 90 | 0.53 (1.25) | 1.40 (1.06) | 2.27 (1.39)
  Day 270 | 0.55 (1.16) | 1.26 (1.53) | 2.30 (1.34)
  Day 365 | 0.88 (1.36) | 0.89 (1.16) | 2.07 (1.23)

8. Secondary Outcome: Number of Subjects With Major, Lower Leg, Amputations During the Trial
Description: The number and percentage of subjects with major amputations during the trial
Time Frame: Day 0 through Day 365
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 11
Participants | 3 | 3 | 1

9. Secondary Outcome: The Number of Deaths During the Trial
Description: The number and percentage of subjects who died during the trial
Time Frame: Day 0 to Day 365
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Engensis (8 mg) | High Dose Engensis (16 mg) | Placebo
Number analyzed (Participants) | 21 | 20 | 11
Participants | 1 | 0 | 1

10. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) for Pain at 9 Months- by Sex
Description: The VAS scoring instrument is a 10 cm line, oriented horizontally, with the left end indicating "no pain" (score = 0 mm, better outcome) and the right end representing "pain as bad as it can be (score = 100 mm, worse outcome).
Time Frame: Days 0 (baseline), 9 months (Day 270)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
Number analyzed (Participants) | 15 | 12 | 5
units on a scale
  Males - Baseline (Day 0) - Actual values only: number analyzed (Participants) | 11 | 6 | 5
  Males - Baseline (Day 0) - Actual values only | 39.1 (31.2) | 70.9 (14.4) | 60.6 (30.1)
  Males - Day 270: number analyzed (Participants) | 11 | 6 | 5
  Males - Day 270 | -6.0 (22.2) | -43.8 (36.2) | -38.6 (41.1)
  Females - Baseline (Day 0) - Actual values only: number analyzed (Participants) | 4 | 6 | 0
  Females - Baseline (Day 0) - Actual values only | 44.3 (36.2) | 53.7 (27.0) |
  Females Day 270: number analyzed (Participants) | 4 | 6 | 0
  Females Day 270 | -14.4 (24.7) | -25.3 (43.9) |

11. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) for Pain at 9 Months- by Renal Dysfunction Status
Description: as for outcome 10
Time Frame: Days 0 (baseline), 9 months (Day 270)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
Number analyzed (Participants) | 15 | 12 | 5
units on a scale
  Has Renal Dysfunction - Baseline (Day 0) - Actual values only: number analyzed (Participants) | 3 | 5 | 2
  Has Renal Dysfunction - Baseline (Day 0) - Actual values only | 13.5 (9.0) | 59.0 (26.8) | 52.0 (38.2)
  Has Renal Dysfunction - Day 270: number analyzed (Participants) | 3 | 5 | 2
  Has Renal Dysfunction - Day 270 | -4.0 (11.1) | -37.1 (45.2) | -27.5 (61.5)
  No Renal Dysfunction - Baseline (Day 0) - Actual values only: number analyzed (Participants) | 12 | 7 | 3
  No Renal Dysfunction - Baseline (Day 0) - Actual values only | 47.2 (31.4) | 64.6 (20.8) | 66.3 (30.9)
  No Renal Dysfunction - Day 270: number analyzed (Participants) | 12 | 7 | 3
  No Renal Dysfunction - Day 270 | -9.3 (24.6) | -32.6 (38.7) | -46.0 (35.7)

12. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) for Pain at 9 Months- by Diabetes Status
Description: as for outcome 10
Time Frame: Days 0 (baseline), 9 months (Day 270)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
Number analyzed (Participants) | 15 | 12 | 5
units on a scale
  Has Diabetes - Baseline (Day 0) - Actual values only: number analyzed (Participants) | 10 | 6 | 2
  Has Diabetes - Baseline (Day 0) - Actual values only | 32.6 (28.0) | 63.8 (21.8) | 77.0 (2.8)
  Has Diabetes - Day 270: number analyzed (Participants) | 10 | 6 | 2
  Has Diabetes - Day 270 | -4.2 (21.3) | -48.2 (29.3) | -46.5 (34.6)
  No Diabetes - Baseline (Day 0) - Actual values only: number analyzed (Participants) | 5 | 6 | 3
  No Diabetes - Baseline (Day 0) - Actual values only | 56.3 (34.8) | 60.8 (25.2) | 49.7 (36.8)
  No Diabetes - Day 270: number analyzed (Participants) | 5 | 6 | 3
  No Diabetes - Day 270 | -16.3 (24.4) | -20.8 (46.3) | -33.3 (51.6)

ADVERSE EVENTS:
Arm/Group | Engensis 8 mg | Engensis 16 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/21 | 0/20 | 1/11
Serious Adverse Events (participants affected / at risk) | 9/21 | 11/20 | 6/11
Other Adverse Events (participants affected / at risk) | 18/21 | 18/20 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis 8 mg (N=21) | Engensis 16 mg (N=20) | Placebo (N=11)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2) | 4 (5) | 1 (2)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 2 (3) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Osteomyelitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 3 (6) | 1 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Arterial stenosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic limb pain (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Celulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 3 (6) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis 8 mg (N=21) | Engensis 16 mg (N=20) | Placebo (N=11)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2) | 2 (3)
Wound infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 2 (10) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Labyrinithitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (4) | 2 (4) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2011-07-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT01064440/Prot_000.pdf
  • Statistical Analysis Plan (2013-10-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT01064440/SAP_001.pdf